CLINICAL TRIAL: NCT01543932
Title: Comparison of Therapy With TICAGRELOR, Prasugrel and High Clopidogrel Dose in PCI Patients With High on Treatment Platelet Reactivity and Genotype Variation
Brief Title: High Clopidogrel Dose Versus Prasugrel and Ticagrelor in High Reactive Stable Patients
Acronym: TRIPLETE RESET
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Gennaro Sardella, Associate Professor in Cardiology, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRIPLETE RESET
Record Dates: First submitted 2012-02-21; First posted 2012-03-05 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Coronary Artery Disease
Keywords: antiplatelet effect; prasugrel; clopidogrel; stable angina
MeSH Terms: conditions — Coronary Artery Disease; Angina, Stable | interventions — Clopidogrel; Prasugrel Hydrochloride; Ticagrelor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Prasugrel standard dose (Experimental): Patient will be randomized to this intervention will receive in the first time prasugrel and after 15 days and 30 days we will control the responsivness of the study drug.
  Interventions: Drug: Prasugrel
- high clopidogrel dose (Experimental): Patient will be randomized to this intervention will receive in the first time the high clopidogrel dose and after 15 days and 30 days we will control the responsivness of the study drug.
  Interventions: Drug: Clopidogrel
- Ticagrelor standard dose (Experimental): Patient will be randomized to this intervention will receive in the first time ticagrelor and after 15 days and 30 days we will control the responsivness of the study drug.
  Interventions: Drug: Ticagrelor

INTERVENTIONS:
Drug: Clopidogrel — Patient will be randomized to this intervention will receive in the first time the double dose of clopidogrel and after 15 days and 30 days we will control the responsivness of the study drug.
  Arms: high clopidogrel dose
Drug: Prasugrel — Patient will be randomized to this intervention will receive in the first time prasugrel and after 15 days and 30 days we will control the responsivness of the study drug.
  Arms: Prasugrel standard dose
Drug: Ticagrelor — Patient will be randomized to this intervention will receive in the first time Ticagrelor and after 14 days and 28 days we will change their therapy with the high clopidogrel dose or Prasugrel (dual crossover).
  Arms: Ticagrelor standard dose

SUMMARY:
Dual antiplatelet therapy with Aspirin and Clopidogrel for at least one year is essential in patients following an acute coronary syndrome (ACS) or percutaneous coronary intervention (PCI) with drug eluting stent(s) implantation. Interindividual variability in platelet response to Clopidogrel has been reported, with several mechanisms (intrinsic high platelet reactivity [PR], variability of the drug metabolism, and various drug interactions) being implicated for high post-Clopidogrel treatment PR. The investigators aim to perform a prospective, single-center, investigator-initiated, randomized, study to compare platelet inhibition by Prasugrel 10 mg/day, Ticagrelor (90 mg twice daily) and high-dose 150 mg/day Clopidogrel in patients with High on-treatment platelet reactivity (HTPR) with standard dose of Clopidogrel. Patients with HTPR (defined as area under curve-AUC ≥ 450 or > 45 Unit) and with loss-of-function allele CYP2C19*2 will be enrolled in the study and will be randomized (Day 0) in a 1:1:1 ratio, to either Clopidogrel 150 mg a day or Prasugrel 10 mg a day or Ticagrelor (90 mg twice daily) until Day-15 and-30 post randomization.

ELIGIBILITY:
Inclusion Criteria:

* patients underwent to percutaneous coronary intervention (PCI)
* clopidogrel resistance after Platelet reactivity blood test

Exclusion Criteria:

* history of bleeding diathesis
* chronic oral anticoagulation treatment
* contraindications to antiplatelet therapy
* PCI or coronary artery bypass grafting (CABG) < 3 months
* hemodynamic instability
* platelet count < 100,000/μl
* hematocrit < 30%
* creatinine clearance < 25 ml/min
* Patients with a history of stroke
* contraindication for prasugrel administration
* patients weighing < 60 kg
* > 75 years of age.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2012-07; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
antiplatelet effect of standard dose of prasugrel or ticagrelor versus high dose clopidogrel in stable patients with high reactivity | 30 days
  the antiplatelet effect in terms of level platelet reactivity (< 450 Area under the curve (AU*min)) of standard dose of Prasugrel (10 mg/day) either Ticagrelor (90 mg twice daily) versus high dose Clopidogrel (150 mg/day) in patients undergoing PCI with high reactivity

SECONDARY OUTCOMES:
Bleeding (major, minor, or minimal) | 45 days
  Bleeding (major, minor, or minimal)
Major Adverse Cardiac Cerebrovascular Events | 45 days
  cardiovascular death, myocardial infarction, and stroke

CONTACTS AND LOCATIONS:
Locations (1):
- Dept.of Cardiovascular Sciences,Policlinico Umberto I, Rome, Rome, Italy

REFERENCES:
- [Derived] Sardella G, Calcagno S, Mancone M, Lucisano L, Pennacchi M, Stio RE, Placentino F, Di Roma A, Cavallo E, Palmirotta R, Guadagni F, Fedele F. Comparison of therapy with Ticagrelor, Prasugrel or high Clopidogrel dose in PCI patients with high on treatment platelet reactivity and genotype variation. TRIPLETE RESET trial. Int J Cardiol. 2015 Sep 1;194:60-2. doi: 10.1016/j.ijcard.2015.05.085. Epub 2015 May 15. No abstract available. PMID 26011265